CLINICAL TRIAL: NCT02601586
Title: Evaluation of the Analgesic Effects of Prolonged-release Oxycodone and of Levodopa, Versus Placebo, on Central Neuropathic Pain in Parkinson's Disease: OXYDOPA Trial
Brief Title: Effects of PR Oxycodone and of Levodopa, vs Placebo, on Central Neuropathic Pain in Parkinson's Disease
Acronym: OXYDOPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14 7440 01
Record Dates: First submitted 2015-08-17; First posted 2015-11-10 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PR oxycodone (Experimental): A titration phase of two weeks, in three steps:
  Level 1 (from D1 to D5):
  * Oxycodone : 10 mg PR/day bid (5 mg PR/5 mg PR)
  * Levodopa placebo 100 mg/day bid (50 mg/50 mg)
  Level 2 (from D6 to D10):
  * Oxycodone : 20 mg PR/day tid (10 mg/0 mg/10 mg)
  * Levodopa placebo: 150 mg/day tid (50 mg/50 mg/50 mg)
  Level 3 (from D11to D15):
  * Oxycodone: 40 mg PR/day tid (20 mg/0 mg/20 mg)
  * Levodopa placebo: 200 mg/day tid (100 mg/50 mg/50 mg)
    * A fixed dose period: the level 3 dose will be maintained for 8 weeks (from D16 to D71).
    * A withdrawal period:
  Interventions: Drug: PR Oxycodone; Drug: Levodopa placebo
- levodopa (Active Comparator): A titration phase of two weeks, in three steps:
  Level 1 (from D1 to D5):
  * Oxycodone placebo : 10 mg PR/day bid (5 mg PR/5 mg PR)
  * Levodopa 100 mg/day bid (50 mg/50 mg)
  Level 2 (from D6 to D10):
  * Oxycodone placebo: 20 mg PR/day tid (10 mg/0 mg/10 mg)
  * Levodopa : 150 mg/day tid (50 mg/50 mg/50 mg)
  Level 3 (from D11to D15):
  * Oxycodone placebo: 40 mg PR/day tid (20 mg/0 mg/20 mg)
  * Levodopa : 200 mg/day tid (100 mg/50 mg/50 mg)
    * A fixed dose period: the level 3 dose will be maintained for 8 weeks (from D16 to D71).
    * A withdrawal period:
  Interventions: Drug: Levodopa; Drug: Oxycodone Placebo
- Placebo (Placebo Comparator): A titration phase of two weeks, in three steps:
  Level 1 (from D1 to D5):
  * Oxycodone placebo : 10 mg PR/day bid (5 mg PR/5 mg PR)
  * Levodopa placebo 100 mg/day bid (50 mg/50 mg)
  Level 2 (from D6 to D10):
  * Oxycodone placebo: 20 mg PR/day tid (10 mg/0 mg/10 mg)
  * Levodopa placebo: 150 mg/day tid (50 mg/50 mg/50 mg)
  Level 3 (from D11to D15):
  * Oxycodone placebo: 40 mg PR/day tid (20 mg/0 mg/20 mg)
  * Levodopa placebo: 200 mg/day tid (100 mg/50 mg/50 mg)
    * A fixed dose period: the level 3 dose will be maintained for 8 weeks (from D16 to D71).
    * A withdrawal period:
  Interventions: Drug: Oxycodone Placebo; Drug: Levodopa placebo

INTERVENTIONS:
Drug: PR Oxycodone — PR Oxycodone
  Other Names: PR Oxycontin
  Arms: PR oxycodone
Drug: Levodopa — Levodopa
  Other Names: Modopar
  Arms: levodopa
Drug: Oxycodone Placebo — Placebo of PR Oxycodone
  Arms: Placebo; levodopa
Drug: Levodopa placebo
  Arms: PR oxycodone; Placebo

SUMMARY:
This study will be conducted in three parallel groups receiving oxycodone, levodopa or placebo, administered as an add-on therapy, in addition to the usual antiparkinsonian treatment. As this study focuses on chronic central neuropathic pain caused by PD, the effects of study treatments will be evaluated after a 10-week treatment period

DETAILED DESCRIPTION:
The treatment period (11 weeks) will be divided into three periods:

1. A titration phase of two weeks, during which of the doses of the treatments will be gradually increased in three steps:

   Level 1 (from D1 to D5):
   * Oxycodone: 10 mg PR/day bid (5 mg PR/5 mg PR)
   * Levodopa: 100 mg/day bid (50 mg/50 mg)

   Level 2 (from D6 to D10):
   * Oxycodone: 20 mg PR/day tid (10 mg/0 mg/10 mg)
   * Levodopa: 150 mg/day tid (50 mg/50 mg/50 mg)

   Level 3 (from D11to D15):
   * Oxycodone: 40 mg PR/day tid (20 mg/0 mg/20 mg)
   * Levodopa: 200 mg/day tid (100 mg/50 mg/50 mg)
2. A fixed dose period: the level 3 dose will be maintained for 8 weeks (from D16 to D71). The study treatment will be administered as an add-on therapy, with the usual antiparkinsonian treatment. If patients have side effects at the level 3 dose, a return to the level 2 dose will be authorized.
3. A withdrawal period: The dose of the study treatment will gradually be reduced, over an eight-day period:

For patients treated with the level 3 dose for 8 weeks: decrease to the level 2 dose over the first 3 days (from D72 to D74) ; then a decrease to the level 1 dose over the next 3 days (from D75 to D77). The treatment will be stopped completely on D78. The last visit will take place on D79, 2 days after the end of treatment.

For patients treated with the level 2 dose: decrease to the level 1 dose over the first 3 days (from D72 to D74), with stopping of the treatment on D75. The last visit will take place on D79, 5 days after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease according to the UKPDSBB (United Kingdom Parkinson's Disease Society Brain Bank) criteria
* Patients suffering from chronic pain (lasting for more than 3 months)
* Patients suffering from central neuropathic pain caused by PD,
* Patients with a PD-related central neuropathic pain intensity of at least 3 points on the VAS (average intensity over the last month),
* Patients with both types of pain (neuropathic and nociceptive) will be included if the neuropathic pain predominates
* Patients treated with a stable regimen of dopaminergic drugs (levodopa and/or dopamine agonists) for at least 4 weeks before the study dan throughout the study
* Patients with a stable step 1 analgesic (NSAIDS, acetaminophen) or coanalgesic (antidepressants, antiepileptic) treatment for at least 4 weeks before the study and throughout the study

Exclusion Criteria:

* Patients suffering from another parkinsonian syndrome
* De Novo patients (patients never before treated with dopaminergic drugs)
* Patients with intercurrent acute pain
* Patients suffering from a chronic disease causing pain (rheumatoid arthritis, ankylosing spondylitis, diabetic neuropathy, cancer etc.)
* Patients treated with neuroleptics
* Patients with clinically detectable behavioural disorders and addiction
* Patients with disabling dyskinesias
* Patients with painful restless legs syndrome
* Patients with cognitive impairment (MMS < 25) or unable to complete the various scales used in the study
* Hypersensitivity to oxycodone, levodopa, benserazide or a combination of these drugs
* Patients treated with opioid drugs (step 2 and 3)
* Patients treated with non-selective monoamine oxidase inhibitors (MAOI)
* Patients with severe hepatocellular insufficiency
* Patients with uncontrolled cardiovascular and pulmonary diseases
* Persistent constipation that has already resulted in a subocclusive state
* Patients treated with antiemetic neuroleptics
* Patients with angle-closure glaucoma

Exclusion criteria relating to MRI:

* Patients with claustrophobia
* Patients with a hearing aid, cardiac prosthesis, pacemaker, surgical clip
* Patients refusing to be informed of abnormalities are detected on MRI

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | 8 weeks
  Change in average pain rated on visual analog scale (VAS) intensity between baseline and after 8 weeks

SECONDARY OUTCOMES:
Maximal pain intensity | 8 weeks
  Change of maximal pain intensity over the preceding week rated on the VAS
Functional impact of pain" of the Brief Pain Inventory (BPI) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Neuropathic Pain Symptoms Inventory (NPSI) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
McGill pain questionnaire (SFMPQ) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Depression and anxiety: the Hospital Depression and Anxiety (HAD) scale | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Apathy: the Lille Apathy Rating Scale (LARS) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Fatigue : the Parkinson fatigue scale | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Sleep : the Pittsburgh sleep quality index | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Motor assessment and motor fluctuations: MDS UPDRS (MDS Movement Disorder Society - UPDRS Unified Parkinson Disease Rating Scale) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Quality of life: Parkinson's Disease Questionnaire 39 items (PDQ-39) | 8 weeks
  Change in scores between Day 0 and Day 71(Day 71= 8 weeks of treatment)
Acetaminophen consumption reported in diary | 8 weeks
  number of pills or capsules reported in patients diary
Adverse events | Day 5, Day 10, Day 15, Day 43, Day 71, Day 79
  Adverse events, evaluated with an open-ended questionnaire
changes in Resting-state brain network (3T fMRI) | Day 0 /Day 71(Day 71= 8 weeks of treatment)
  changes in resting-state cerebral networks between Day 0 and Day 71, as assessed by 3T fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, MD, Principal Investigator — University Hospital, Toulouse; Claire THALAMAS, MD, Study Chair — University Hospital, Toulouse
Locations (18):
- France (18):
  - Hospital of Aix-en-Provence, Aix-en-Provence
  - CHU Amiens, Amiens
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - Henri Mondor Hospital, Créteil
  - University Hospital of Lille, Lille
  - University Hospital of Limoges, Limoges
  - Hospital Pierre Wertheimer, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nîmes - Caremeau, Nîmes
  - Pitié-Salpêtrière Hospital, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse

REFERENCES:
- [Derived] Lawn T, Rukavina K, Malcangio M, Howard M, Chaudhuri KR. Response to Mylius et al. Pain. 2022 Mar 1;163(3):e496-e497. doi: 10.1097/j.pain.0000000000002445. No abstract available. PMID 35148289